CLINICAL TRIAL: NCT01077232
Title: Long Term Documentation of the Safety and Efficacy as Well as the Effects on Work Productivity in Patients With Moderate to Severe Plaque Psoriasis Treated With HUMIRA (Adalimumab) in Routine Clinical Practice (LOTOS)
Brief Title: Documentation of Humira in Psoriasis Patients in Routine Clinical Practice
Acronym: LOTOS
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P10-446
Record Dates: First submitted 2010-02-25; First posted 2010-03-01 (Estimated); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Moderate to Severe Plaque Psoriasis
Keywords: Moderate to Severe Plaque Psoriasis; Humira; Safety; Efficacy; Work Productivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Psoriasis Patients: Patients with moderate to severe plaque psoriasis

SUMMARY:
Safety and Effectiveness of adalimumab (Humira) in Psoriasis Patients in Routine Clinical Practice.

DETAILED DESCRIPTION:
Postmarketing Observational Study to Evaluate the Work Productivity, Safety and Efficacy of Humira for the Treatment of Moderate to Severe Plaque Psoriasis in Daily Clinical Practice. The primary objectives of the PMOS are to explore changes in health related care utilization data by the evaluation of:

* the number of missed working days
* the number of visits to doctor's office
* the number and duration of hospitalizations
* work ability to assess efficacy for different subgroups by
* the number of patients achieving a PASI 75 response to evaluate safety by
* the documentation and analysis of adverse events for all patients and subgroups with concomitant diseases Secondary objectives include the exploration of changes in quality of life measurements, of the influence of age, gender and duration of disease

ELIGIBILITY:
Inclusion Criteria:

- Moderate to severe plaque psoriasis in adults with no response to other systemic therapy (e.g. cyclosporine, methotrexate or PUVA (photochemical therapy)) or patients with a contraindication or hypersensitivity to such a therapy

Exclusion Criteria:

- Hypersensitivity against the drug or one of the other ingredients; active tuberculosis or other severe infections (e.g. sepsis and opportunistic infections); moderate to severe cardiac insufficiency

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community Sample: Patients with Plaque Psoriasis
Sampling Method: Non-Probability Sample
Enrollment: 5442 (Actual)
Dates: Start 2008-01-04 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in Psoriasis Area and Severity Index; number of patients with Psoriasis Area and Severity Index-75 reduction. | At 24, 48 and 60 months
Changes in healthcare parameters: number of missed working days due to psoriasis; number of visits at the doctor's office; number and duration of hospitalizations, self-assessed workability. | At 24, 48 and 60 months
Safety and tolerability assessed by analyzing serious and non-serous adverse events. | At 24, 48 and 60 months

SECONDARY OUTCOMES:
Global physician's assessment on Humira treatment. | At 24, 48 and 60 months
Target Nail Psoriasis Severity Index (target NAPSI). | At 24 months
Itch Visual Analogue Scale (Itch VAS). | At 24 months
Safety and tolerability of Humira - treatment for patient groups with frequent concommitant diseases, especially diabetes type I and II, cardio-vascular and liver and kidney functional impairment and respective concommitant medication. | At 24, 48 and 60 months
Palmoplantar Psoriasis Area Severity Index (pPASI). | At 24 months
Influence of body mass index and weight on efficacy measurement. | At 24, 48 and 60 months
Patients' assessment on Humira treatment. | At 24, 48 and 60 months

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (641):
- Germany (641):
  - Universitaetsklinik Heidelberg /ID# 33810, Heidelberg, Baden-Wurttemberg
  - Universitaetsklinik Heidelberg /ID# 50858, Heidelberg, Baden-Wurttemberg
  - Universitatsklinikum Mannheim /ID# 166130, Mannheim, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen /ID# 34816, Erlangen, Bavaria
  - Universitätsklinikum Frankfurt /ID# 53725, Frankfurt am Main, Hesse
  - Universitatsklinikum Munster /ID# 205840, Munster, Lower Saxony
  - Universitatsklinikum Munster /ID# 72018, Munster, Lower Saxony
  - Universitatsklinikum Munster /ID# 72022, Munster, Lower Saxony
  - Praxis M. Vilic /ID# 210108, Aachen, North Rhine-Westphalia
  - Universitaetsklinikum Aachen /ID# 35037, Aachen, North Rhine-Westphalia
  - Uniklinik Koln /ID# 166128, Cologne, North Rhine-Westphalia
  - Hautarztpraxis am Buddenturm /ID# 205094, Münster, North Rhine-Westphalia
  - Praxis Dr. Büchner /ID# 204352, Dresden, Saxony
  - Universitaetsklinikum Leipzig /ID# 53720, Leipzig, Saxony
  - Praxis Dr. Reimann /ID# 142004, Pirna, Saxony
  - Praxis N. Yenigün /ID# 206670, Kiel, Schleswig-Holstein
  - Univ Hosp Schleswig-Holstein /ID# 33981, Kiel, Schleswig-Holstein
  - Univ Hosp Schleswig-Holstein /ID# 35269, Kiel, Schleswig-Holstein
  - Medizinisches Versorgungszentrum DermaKiel GmbH /ID# 33972, Kiel, Schleswig-Holstein
  - Hoeller-Obrigkeit, Aachen, DE /ID# 60599, Aachen
  - Petri, Ahaus, DE /ID# 53712, Ahaus
  - Gewiss, Ahrensburg, DE /ID# 33431, Ahrensburg
  - Praxis Dr. Schuessler /ID# 149404, Alsfeld
  - Oster-Schmidt, Altenkirchen, D /ID# 126022, Altenkirchen
  - Weiss, Amberg, DE /ID# 60613, Amberg
  - Dietz, Ampfing, DE /ID# 50790, Ampfing
  - Bell, Andernach, DE /ID# 99815, Andernach
  - Schulz, Angermuende, DE /ID# 53719, Angermünde
  - Rebbien, Annaberg-Buchholz, DE /ID# 35052, Annaberg-Buchholz
  - Thieme, Artern, DE /ID# 35518, Artern
  - Dr. Szlava Fuezesi, Achaffenbu /ID# 118537, Aschaffenburg
  - Theuring, Aschersleben, DE /ID# 35058, Aschersleben
  - Hums, Aue, DE /ID# 60601, Aue
  - Gerloff-Steiner, Aue, DE /ID# 53694, Aue
  - Schneider & Sedlmayr, Augsburg /ID# 33351, Augsburg
  - Lechner/Stuebich, Aurich, DE /ID# 33355, Aurich
  - Lechner/Stuebich, Aurich, DE /ID# 67967, Aurich
  - Brautzsch, Bad Berka, DE /ID# 33365, Bad Berka
  - Broschewitz/Hammer Bad Doberan /ID# 60596, Bad Doberan
  - Broschewitz/Hammer Bad Doberan /ID# 67948, Bad Doberan
  - Mauer, Bad Kreuznach, DE /ID# 126019, Bad Kreuznach
  - Schulz, Bad Muender, DE /ID# 48469, Bad Münder am Deister
  - SALUS-Klinik /ID# 33405, Bad Reichenhall
  - Praxis Dr. Bock /ID# 166127, Bad Rothenfelde
  - Houda, Bad Schlema, DE /ID# 35584, Bad Schlema
  - Moerstedt, Bad Woerishofen, DE /ID# 99844, Bad Wörishofen
  - Sozialstiftung Bamberg /ID# 33430, Bamberg
  - Stephan-Dahm, Bargteheide, DE /ID# 50861, Bargteheide
  - Dr. Roxana Homolka, Baunatal, /ID# 118539, Baunatal
  - Mirtschink, Bautzen, DE /ID# 50851, Bautzen
  - Graessel, Bayreuth, DE /ID# 35587, Bayreuth
  - Kinateder, Bayreuth, DE /ID# 33439, Bayreuth
  - Blaese & Walther, Bendorf, DE /ID# 50787, Bendorf
  - Pflieger-Bruss, Benndorf, DE /ID# 53713, Benndorf
  - Timmel/Timm/Vorwerk, Bergen /ID# 33451, Bergen
  - Wirtler, Bergisch Gladbach, DE /ID# 33452, Bergisch Gladbach
  - Charité Universitätsmedizin Campus Mitte /ID# 33457, Berlin
  - Hasert & Hasert, Berlin, DE /ID# 35531, Berlin
  - Kindler, Berlin, Germany /ID# 60604, Berlin
  - Klusmann, Berlin, DE /ID# 90974, Berlin
  - Spickermann, Berlin, DE /ID# 33675, Berlin
  - Praxis Dermatologie am Savigny /ID# 145783, Berlin
  - Herzler & Reupke, Berlin, DE /ID# 33705, Berlin
  - Boodstein, Berlin, Germany /ID# 48417, Berlin
  - Rothhaar, Berlin, DE /ID# 33644, Berlin
  - Simon, Berlin, DE /ID# 33678, Berlin
  - Steinhoff-Georgieva, Berlin,DE /ID# 60612, Berlin
  - Struss, Berlin, DE /ID# 33680, Berlin
  - Miller/Nerenheim, Berlin, DE /ID# 99842, Berlin
  - Praxis Dr. med. Meljanac /ID# 151477, Berlin
  - Praxis Dr. med. Meljanac /ID# 35594, Berlin
  - Jacob, Berlin, DE /ID# 48438, Berlin
  - Vivantes Klinikum Neukolln /ID# 34270, Berlin
  - Weihe/Stavermann, Berlin, DE /ID# 35547, Berlin
  - Gellrich, Berlin, DE /ID# 33691, Berlin
  - Schirmer, Berlin, DE /ID# 35534, Berlin
  - Skarabis/Skarabis, Berlin, DE /ID# 34241, Berlin
  - Kv Be /Id# 34253, Berlin
  - Praxis Dres. Eicholtz/Boerner /ID# 167676, Berlin
  - Wildfeuer, Berlin, DE /ID# 33694, Berlin
  - Kors, Berlin, DE /ID# 33649, Berlin
  - Zahn, Berlin, DE /ID# 35592, Berlin
  - Praxis Dr. Uhl /ID# 171308, Berlin
  - Dues/Manasterski, Berlin, DE /ID# 35538, Berlin
  - Miehe & Partner, Berlin, DE /ID# 166125, Berlin
  - Miehe & Partner, Berlin, DE /ID# 35544, Berlin
  - Baumann, Berlin, DE /ID# 60584, Berlin
  - Groene, Berlin, DE /ID# 60594, Berlin
  - Neumann, Bernau, DE /ID# 34271, Bernau
  - Praxis Dr. Duhn /ID# 167672, Bernau bei Berlin
  - Biel, Bielefeld, DE /ID# 60586, Bielefeld
  - MVZ Otto-Brenner-Straße /ID# 167677, Bielefeld
  - Staedt Kliniken Bielefeld /ID# 35558, Bielefeld
  - Dabour & Dabour, Birkenwerder /ID# 34280, Birkenwerder
  - Wege & Kuehnast, Bitterfeld /ID# 34282, Bitterfeld-Wolfen
  - Praxis fuer Innere Medizin/Rhe /ID# 35564, Blaubeuren Abbey
  - Ruppert, Bocholt, DE /ID# 108918, Bocholt
  - Klinikum Ruhr Univ Bochum /ID# 35091, Bochum
  - GP Dr. Niesman & Dr. Othlingha /ID# 169694, Bochum
  - Ardabili/Niesmann, Bochum, DE /ID# 50784, Bochum
  - Universitaetsklinikum Bonn /ID# 34299, Bonn
  - Praxis Dr. Schift /ID# 141549, Borken
  - Barth, Borna, DE /ID# 35650, Borna
  - Barth, Borna, DE /ID# 67946, Borna
  - Alte Apotheke /ID# 48530, Bottrop
  - Flont-Schmeling, Bottrop, DE /ID# 48423, Bottrop
  - Karpinski, Bottrop, DE /ID# 34303, Bottrop
  - Tolzin, Brake, DE /ID# 50866, Brake
  - Praxis S. Osadtschy /ID# 161167, Brandenburg
  - Klee/Wolff, Brandenburg, DE /ID# 67960, Brandenburg
  - Atugoda, Braunschweig, DE /ID# 48509, Braunschweig
  - Gaedt, Braunschweig, DE /ID# 67954, Braunschweig
  - Koehn & Ramaker-Brunke, DE /ID# 34309, Braunschweig
  - Klinikverbund Bremen /ID# 171306, Bremen
  - Elsner, Bremen, DE /ID# 48422, Bremen
  - Derma am Diako /ID# 166131, Bremen
  - Hermann/Teichelmann, Bremen,DE /ID# 35605, Bremen
  - Altvater/Tauschke, Bremen, DE /ID# 34311, Bremen
  - Schwichtenberg, Bremen, DE /ID# 34312, Bremen
  - Friedmann, Bremerhaven, DE /ID# 67952, Bremerhaven
  - Heitmann, Bremerhaven, DE /ID# 148410, Bremerhaven
  - Bessle, Buchholz, DE /ID# 60585, Buchholz
  - Streit, Buchholz, DE /ID# 53723, Buchholz I.D. Nordheide
  - Arensmeier-Gottschalkson, Burg /ID# 48508, Burg
  - Praxis K. Neubert /ID# 149400, Burgstädt
  - Wagenpfeil, Burscheid, DE /ID# 99856, Burscheid
  - Elbe Klinikum Buxtehude /ID# 34694, Buxtehude
  - Praxis B. Jaeckel /ID# 145768, Chemnitz
  - Jaeckel & Partner, Chemnitz, D /ID# 34703, Chemnitz
  - Kuehn/Stengel, Chemnitz, DE /ID# 90978, Chemnitz
  - Praxis P. Hausler-Mehlhorn /ID# 149285, Chemnitz
  - Schneider, Chemnitz, DE /ID# 35613, Chemnitz
  - Hoffmann, Coburg, DE /ID# 34704, Coburg
  - Pappai, Coesfeld, DE /ID# 108917, Coesfeld
  - Karger/Rezazadegan, Cologne DE /ID# 60608, Cologne
  - Menge & Franckson, Cologne, DE /ID# 53708, Cologne
  - Haitas-Haase, Cologne, DE /ID# 53696, Cologne
  - Haase & Partner, Cologne, DE /ID# 53724, Cologne
  - Praxis Dres. Neuhaus/Sacha /ID# 149403, Cologne
  - Matias-Bako/Krickeberg,Cologne /ID# 90975, Cologne
  - Eichhorn, Cologne, DE /ID# 99818, Cologne
  - Krebs, Coswig, DE /ID# 48519, Coswig
  - Praxis S.-K. Strenzke /ID# 145781, Cottbus
  - Dr. Bernd Jantsch, Cottbus, DE /ID# 35618, Cottbus
  - Loessner, Cottbus, DE /ID# 34712, Cottbus
  - Dr. Susanne Jantsch,Cottbus,DE /ID# 35619, Cottbus
  - Klinikum Darmstadt GmbH /ID# 34720, Darmstadt
  - Buelow, Delmenhorst, DE /ID# 35626, Delmenhorst
  - Thelen, Delmenhorst, DE /ID# 35628, Delmenhorst
  - Heidlas, Dessau-Rosslau, DE /ID# 34730, Dessau
  - Klinikum Lippe Detmold GmbH /ID# 34731, Detmold
  - Friedrich, Dieburg, DE /ID# 53693, Dieburg
  - Gerharz, Diez, DE /ID# 48432, Diez
  - Winter, Dinkelsbuehl, DE /ID# 34734, Dinkelsbühl
  - Ghassem-Zadeh/Farashahi /ID# 138188, Dormagen
  - Thomas, Dorsten, DE /ID# 34736, Dorsten
  - Brinkmeier & Partner, Dortmund /ID# 138259, Dortmund
  - Brinkmeier & Partner, Dortmund /ID# 99847, Dortmund
  - Hautklinik Dortmund /ID# 72019, Dortmund
  - Hirschmueller, Dortmund, DE /ID# 34737, Dortmund
  - Bebnowski, Dortmund, DE /ID# 53684, Dortmund
  - Dick/Hubert/Mirkin, Dortmund /ID# 99843, Dortmund
  - Frolova, Dortmund, DE /ID# 51022, Dortmund
  - Frach/Hohaus, Dresden, DE /ID# 35166, Dresden
  - Frach/Hohaus, Dresden, DE /ID# 60600, Dresden
  - Gerlach, Dresden, DE /ID# 48433, Dresden
  - Praxis Dres. Pollack Schramm /ID# 149286, Dresden
  - Kuehn, Dresden, DE /ID# 34752, Dresden
  - Schamfuss, Dresden, DE /ID# 48468, Dresden
  - Richter-Huhn, Dresden, DE /ID# 35164, Dresden
  - Hass, Dresden, Germany /ID# 60597, Dresden
  - Meier, Dresden, DE /ID# 48452, Dresden
  - Universitaetklinikum Dresden /ID# 34764, Dresden
  - University Clinic Carl Gustav /ID# 99820, Dresden
  - Praxis Dr. Mayer /ID# 148243, Dresden
  - Scheibner, Dresden, DE /ID# 35162, Dresden
  - Oppers, Dresden, DE /ID# 126021, Dresden
  - Siebert, Duisburg, DE /ID# 34775, Duisburg
  - St. Barbara-Hospital /ID# 81302, Duisburg
  - Praxis. Y. Teoman /ID# 142005, Duisburg
  - Elsner, Duisburg, DE /ID# 99819, Duisburg
  - Saget & Riesopp, Duisburg, DE /ID# 35175, Duisburg
  - Praxis Dr. Lobert /ID# 145774, Duisburg
  - Bockhorst & Dominicus, Duelmen /ID# 34765, Dülmen
  - Korge, Dueren, DE /ID# 35174, Düren
  - Evangelisches Krankenhaus Dues /ID# 48419, Düsseldorf
  - Berendt, Eberswalde, DE /ID# 35178, Eberswalde
  - Badura, Eilenburg, DE /ID# 35179, Eilenburg
  - Praxis Dr. Kues /ID# 145771, Einbeck
  - Dove, Eisenach, DE /ID# 48420, Eisenach
  - Reinhardt, Eisenach, DE /ID# 48465, Eisenach
  - Rast, Eisenhuettenstadt, DE /ID# 34789, Eisenhüttenstadt
  - Richter/Cyw, Eisenhuettenstadt /ID# 34790, Eisenhüttenstadt
  - Noack, Lutherstadt Eisleben,DE /ID# 48521, Eisleben Lutherstadt
  - Schmid, Ellwangen, DE /ID# 34792, Ellwangen
  - Praxis Dr. Fitz /ID# 145767, Elmshorn
  - Hartl, Eltville, DE /ID# 34796, Eltville
  - Med X Aerzteteam GmbH /ID# 90977, Emden
  - Meinert, Emden, DE /ID# 34797, Emden
  - Maurer & Krebs-Posingies /ID# 34800, Emsdetten
  - Schurhammer-Fuhrmann, Endingen /ID# 67966, Endingen
  - Koenig, Erfurg, DE /ID# 99838, Erfurt
  - Nennstiel, Erfurt, DE /ID# 34804, Erfurt
  - Lichtenstein, Eschweiler, DE /ID# 50842, Eschweiler
  - Praxis Dres. Exner/Kanja /ID# 145769, Essen
  - Universitaetsklinikum Essen /ID# 34827, Essen
  - Universitaetsklinikum Essen /ID# 53718, Essen
  - Klundt, Essen, DE /ID# 138195, Essen
  - Praxis Dres. Beyer /ID# 141989, Essen
  - Praxis Dres. Beyer /ID# 90957, Essen
  - Praxis Dr. Porwollik /ID# 148244, Essen
  - Praxis Dres. Renner/Sohl /ID# 149289, Esslingen am Neckar
  - Huerkamp, Euskirchen, DE /ID# 48517, Euskirchen
  - Swirski, Euskirchen, DE /ID# 81314, Euskirchen
  - Praxis Dres. Freitag/Knoell /ID# 167675, Falkensee
  - Jovic-Paris, Bad Neuenahr /ID# 48439, Fitzroy
  - Godt, Flensburg, DE /ID# 67957, Flensburg
  - Praxis T. Zimmermann /ID# 145784, Flöha
  - Eichinger, Frankenberg, DE /ID# 138260, Frankenberg
  - Schoengen/Schwarzenbach, Frank /ID# 60610, Frankenthal
  - Schoengen/Schwarzenbach, Frank /ID# 60611, Frankenthal
  - Kaufmann, Frankfurt, DE /ID# 35098, Frankfurt
  - Hundgeburth, Frechen, DE /ID# 138192, Frechen
  - Kaemmerer, Freiberg, DE /ID# 138194, Freiberg
  - Trefzer, Freiburg im Breisgau, /ID# 126028, Freiburg im Breisgau
  - Kurzen, Freising, DE /ID# 67964, Freising
  - Schmidt, Fuerstenwalde, DE /ID# 34868, Fürstenwalde
  - Gall, Fuerth, DE /ID# 48431, Fürth
  - Teichler, Gaggenau, DE /ID# 99855, Gaggenau
  - Wolf, Garbsen, DE /ID# 99859, Garbsen
  - Praxis Dr. Billmann-Krutmann /ID# 149399, Geilenkirchen
  - Praxis Dres. Kobus / Wetz /ID# 169692, Gelsenkirchen
  - Praxis K. R. Koerber & Partner /ID# 151715, Gelsenkirchen
  - Wetz, Gelsenkirchen, DE /ID# 99858, Gelsenkirchen
  - Rotterdam, Gelsenkirchen, DE /ID# 50856, Gelsenkirchen
  - Praxis J. Teichmann & Partner /ID# 145775, Gelsenkirchen
  - Lange, Dietrich & Beyer, Gera /ID# 48449, Gera
  - Lange, Dietrich & Beyer, Gera /ID# 81274, Gera
  - Paul/Meyer, Gera, DE /ID# 54379, Gera
  - SRH Wald-Klinikum Gera GmbH /ID# 60602, Gera
  - Schnee, Gera, DE /ID# 81313, Gera
  - Estel, Gera, DE /ID# 35226, Gera
  - Loth, Gernsbach, DE /ID# 50844, Gernsbach
  - Gross/Braeu, Giessen, DE /ID# 34884, Giessen
  - Kloevekorn & Tepe, Gilching /ID# 118541, Gilching
  - Kloevekorn & Tepe, Gilching /ID# 48504, Gilching
  - Kloevekorn & Tepe, Gilching /ID# 48506, Gilching
  - Brinkmann & Partner, Gladbeck, /ID# 34889, Gladbeck
  - Brinkmann & Partner, Gladbeck, /ID# 53688, Gladbeck
  - Jahn, Glauchau, DE /ID# 35230, Glauchau
  - Hille, Goerlitz, DE /ID# 60598, Görlitz
  - Cleffmann/Ranke, Goettingen DE /ID# 53689, Göttingen
  - Univ Medical Center Goettingen /ID# 35103, Göttingen
  - Kisslinger/Kisslinger, Grafena /ID# 34897, Grafenau
  - Kuckert, Graefenhainichen, DE /ID# 48520, Gräfenhainichen
  - Herrmann, Greifswald, DE /ID# 72016, Greifswald
  - Manke, Grevesmuehlen, DE /ID# 34907, Grevesmühlen
  - Wigbels, Gronau, DE /ID# 48505, Gronau
  - Grossmann, Grossenhain, DE /ID# 126016, Großenhain
  - Westphal, Guestrow, DE /ID# 35500, Güstrow
  - Busse-Misic, Hagen, DE /ID# 34914, Hagen
  - Timtschenko, Hagen, DE /ID# 138203, Hagen
  - Stehl, Haiger, DE /ID# 126027, Haiger
  - Gstoettner, Halle, DE /ID# 48513, Halle
  - Hamm, Halle, DE /ID# 72015, Halle
  - Lutze, Halle, DE /ID# 34919, Halle
  - Reiss, Halle, DE /ID# 35507, Halle
  - Zarzour, Halle, DE /ID# 35505, Halle
  - Hetschko, Halle, DE /ID# 48437, Halle
  - Universitatsklinikum Halle /ID# 34941, Halle
  - Gagu-Koll, Hamburg, DE /ID# 48424, Hamburg
  - Univ Klinik Eppendorf Hamburg /ID# 35115, Hamburg
  - Univ Klinik Eppendorf Hamburg /ID# 48453, Hamburg
  - Dermatologikum Hamburg /ID# 35107, Hamburg
  - Wagner, Hamburg, DE /ID# 99857, Hamburg
  - Mengert/Nienstedt, Hamburg, DE /ID# 34995, Hamburg
  - Luetten, Hamburg, DE /ID# 50847, Hamburg
  - Kahle/Ohnemus, Hamburg, DE /ID# 148412, Hamburg
  - Praxis Dres. Harms/Hartmann /ID# 148249, Hamburg
  - Buerger, Hamburg, DE /ID# 34966, Hamburg
  - Montag, Hamburg, DE /ID# 35438, Hamburg
  - Buck, Hamburg, DE /ID# 34964, Hamburg
  - Dermatologisches Ambulatorium /ID# 35435, Hamburg
  - Dermatologisches Ambulatorium /ID# 35436, Hamburg
  - Kunze, Hamburg, DE /ID# 34949, Hamburg
  - Kuwert/Wendt/Schulz, Hamburg, /ID# 34991, Hamburg
  - Hautarztpraxis am Tibarg /ID# 35004, Hamburg
  - Schmolke, Hamburg, DE /ID# 67965, Hamburg
  - Wrage-Brors, Hamburg, DE /ID# 126030, Hamburg
  - Szabo, Hamm, DE /ID# 35015, Hamm
  - Weitzel, Hamm, DE /ID# 90982, Hamm
  - Klinikum Hanau gGmbH /ID# 35020, Hanau
  - Praxis U. Stein /ID# 171307, Hanover
  - Theuerkauf, Hanover, DE /ID# 35454, Hanover
  - Stein, Hanover, DE /ID# 35029, Hanover
  - Horstmann, Hanover, DE /ID# 35026, Hanover
  - Durani & Durani, Heidelberg,DE /ID# 48421, Heidelberg
  - Alheit, Heidenau, DE /ID# 50782, Heidenau
  - Pawlak, Heilbad Heiligenstadt, /ID# 138191, Heilbad Heiligenstadt
  - Pawlak, Heilbad Heiligenstadt, /ID# 35466, Heilbad Heiligenstadt
  - Arnold/Kaschubowski/Salzer/Wur /ID# 67971, Heilbronn
  - Arnold/Kaschubowski/Salzer/Wur /ID# 99837, Heilbronn
  - Schulte/Mainusch, Heiligenhaus /ID# 138202, Heiligenhaus
  - Postrach, Hennigsdorf, DE /ID# 35468, Hennigsdorf
  - Praxis G. Taesler /ID# 145782, Herrnhut
  - Allmacher, Hersbruck, DE /ID# 125998, Hersbruck
  - PsoriSol Hautklinik GmbH /ID# 169690, Hersbruck
  - Kroemer, Herten, DE /ID# 48448, Herten
  - Badacz, Heusenstamm, DE /ID# 125999, Heusenstamm
  - Biedenkapp, Heusenstamm, DE /ID# 81275, Heusenstamm
  - Stark & Stark, Hilden, DE /ID# 35470, Hilden
  - Klinken, Hilden, DE /ID# 33829, Hilden
  - Kubek, Hofgeismar, DE /ID# 67963, Hofgeismar
  - Lenz, Hofheim, DE /ID# 33839, Hofheim
  - Praxis Dr. Brill /ID# 145764, Hofheim am Taunus
  - Reinecke, Holzminden, DE /ID# 48464, Holzminden
  - Franke, Homburg, DE /ID# 99821, Homburg
  - Univ Kliniken des Saarlandes /ID# 33848, Homburg
  - Nawka, Pistrosch, Hoyerswerda /ID# 81299, Hoyerswerda
  - Wolz/Bierbaum, Hoyerswerda, DE /ID# 48531, Hoyerswerda
  - Christoph, Ilmenau, DE /ID# 67949, Ilmenau
  - Lutz, Ingolstadt, DE /ID# 35477, Ingolstadt
  - Stockmeier, Ingoldstadt, DE /ID# 53722, Ingolstadt
  - Tuttner, Ingoldstadt, DE /ID# 53726, Ingolstadt
  - Gfesser, Ingolstadt, DE /ID# 81277, Ingolstadt
  - Pueschel, Ingolstadt, DE /ID# 33859, Ingolstadt
  - Universitaetsklinikum Jena /ID# 138198, Jena
  - Brilon & Zanker, Juelich, DE /ID# 33943, Jülich
  - Brilon & Zanker, Juelich, DE /ID# 60614, Jülich
  - Gaehtgens, Kamen, DE /ID# 67955, Kamen
  - Thomas & Heike Mauer,Kamenz,DE /ID# 35480, Kamenz
  - Dres. Bettinger & Kollegen /ID# 138185, Karlsruhe
  - Meyer-Rogge & Kollegen /ID# 72013, Karlsruhe
  - Meyer-Rogge & Kollegen /ID# 99841, Karlsruhe
  - Reitenbach-Blindt,Karlsruhe,DE /ID# 48466, Karlsruhe
  - Glutsch, Karlsruhe, DE /ID# 33953, Karlsruhe
  - Eichbauer, Karlsruhe, DE /ID# 126017, Karlsruhe
  - Eichbauer, Karlsruhe, DE /ID# 60592, Karlsruhe
  - Dunkel, Karlstadt, DE /ID# 50822, Karlstadt am Main
  - Fueller, Kassel, DE /ID# 67953, Kassel
  - Medikum MVZ GmbH /ID# 148248, Kassel
  - Meyer & Baum, Kassel, DE /ID# 108916, Kassel
  - Meyer & Baum, Kassel, DE /ID# 50785, Kassel
  - Kreiselmaier, Kiel, DE /ID# 81298, Kiel
  - Klee/Radeck, Kleinmachnow, DE /ID# 33982, Kleinmachnow
  - Giesen, Kleve, DE /ID# 50825, Kleve
  - Grosse, Kleve, DE /ID# 33983, Kleve
  - Grossmann, Koblenz, DE /ID# 99835, Koblenz
  - Habermann, Koblenz, DE /ID# 35488, Koblenz
  - Blisse, Koenigs Wusterhausen, /ID# 33999, Königs Wusterhausen
  - Gruner, Koenigs Wusterhausen, /ID# 33998, Königs Wusterhausen
  - Hetzer/Schuster/Prothmann /ID# 138200, Krefeld
  - Hetzer/Schuster/Prothmann /ID# 50860, Krefeld
  - Gerhards, Krefeld, DE /ID# 108915, Krefeld
  - Sauer/Wolff/Kreiss, Krefeld, D /ID# 141546, Krefeld
  - Sauer/Wolff/Kreiss, Krefeld, D /ID# 35242, Krefeld
  - Sauer/Wolff/Kreiss, Krefeld, D /ID# 53705, Krefeld
  - Praxis Dres. Hartschuh/Sugar-B /ID# 167674, Krumbach
  - Sugar-Bunk, Krumbach, DE /ID# 34085, Krumbach
  - Dres. Jacobs & Kollegen /ID# 149402, Kulmbach
  - Schmidt, Kusel, DE /ID# 60609, Kusel
  - Fritz/Biwer/Scherer/Uhlig /ID# 149401, Landau
  - Huppmann, Landshut, DE /ID# 72017, Landshut
  - Jacoby, Landshut, DE /ID# 34089, Landshut
  - Janecka, Langenfeld, DE /ID# 34090, Langenfeld
  - Glockemann/Vennemann, Langenha /ID# 34091, Langenhagen
  - Glockemann/Vennemann, Langenha /ID# 53728, Langenhagen
  - Praxis. C. Nitzschner /ID# 142001, Langenselbold
  - Praxis Dr. Juttner /ID# 169691, Lauda-Königshofen
  - Riebel & Meckl & Goetz, Lauf /ID# 34093, Lauf
  - Schunter, Laupheim, DE /ID# 35247, Laupheim
  - Biedermann-Hahn, Lauterbach,DE /ID# 48416, Lauterbach
  - Wirbel, Lehrte, DE /ID# 53730, Lehrte
  - Noack-Wiemers, Leipzig, DE /ID# 35248, Leipzig
  - Gruenenwald, Leipzig, DE /ID# 60595, Leipzig
  - Neubauer, Leipzig, DE /ID# 34103, Leipzig
  - Adler, Lengenfeld, DE /ID# 34115, Lengenfeld
  - Ogger & Gueldner-Engelmann /ID# 48455, Leonberg
  - Onsa, Leverkusen, DE /ID# 90976, Leverkusen
  - Praxis Dr. Carl /ID# 148247, Lichtenfels
  - Dielmann, Limburg, DE /ID# 34124, Limburg
  - Vehring/Amann/Beier,Lingen,DE /ID# 35251, Lingen
  - Schuermeyer-Horst, Lippstadt, /ID# 34126, Lippstadt
  - Grodzki & Pier, Lippstadt, DE /ID# 34128, Lippstadt
  - Grodzki & Pier, Lippstadt, DE /ID# 48523, Lippstadt
  - Lochno, Loebau, DE /ID# 50843, Löbau
  - Hagemeier, Loehne, DE /ID# 35256, Löhne
  - Ifflaender, Luckenwalde, DE /ID# 50828, Luckenwalde
  - Schultz, Ludwigsfelde, DE /ID# 50859, Ludwigsfelde
  - Boehm & Boehm, Ludwigshafen /ID# 35263, Ludwigshafen
  - Wiest/Meng, Ludwigshafen, DE /ID# 138196, Ludwigshafen
  - Klinikum Stadt Ludwigshafen/Rh /ID# 34131, Ludwigshafen
  - Kreusch/Krengel/Mrowka, Luebec /ID# 148411, Lübeck
  - Thierfelder, Luebeck, DE /ID# 34132, Lübeck
  - Dlugosz-Wolf, Luedenscheid, DE /ID# 81276, Lüdenscheid
  - Praxis Dr. Bause /ID# 167670, Lüdenscheid
  - Maerkische Kliniken GmbH /ID# 48512, Lüdenscheid
  - Praxis Ch. Nolting-Schraeer /ID# 141548, Lüdinghausen
  - Birkner-Porath, Lueneburg, DE /ID# 90959, Lüneburg
  - Praxis C. Besser /ID# 141988, Lünen
  - Bruecher, Magdeburg, DE /ID# 126000, Magdeburg
  - Grasshoff, Magdeburg, DE /ID# 34144, Magdeburg
  - Praxis Dr. Kuehne /ID# 145773, Magdeburg
  - Genseke/Krause, Magdeburg, DE /ID# 149288, Magdeburg
  - Kuchheuser, Magdeburg, DE /ID# 34143, Magdeburg
  - Otto von Guericke Universitaet /ID# 48435, Magdeburg
  - Otto von Guericke Universitaet /ID# 60588, Magdeburg
  - Drs Scholz/Sebastian/Schilling /ID# 35273, Mahlow
  - Univ Johannes Gutenberg /ID# 35662, Mainz
  - Knuechel, Mannheim, DE /ID# 48440, Mannheim
  - Richter & Schernitzky,Mannheim /ID# 34183, Mannheim
  - Fuchs, Markdorf, DE /ID# 90973, Markdorf
  - Schulze/Schulze, Markkleeberg, /ID# 34188, Markkleeberg
  - Maassen, Maxdorf, DE /ID# 34197, Maxdorf
  - Cymorek, Meinerzhagen, DE /ID# 48511, Meinerzhagen
  - Werner, Meissen, DE /ID# 81318, Meissen
  - Schwinn & Winkler,Memmingen,DE /ID# 35281, Memmingen
  - Moeller-Massling & Wippermann /ID# 48529, Menden
  - Klinikum Minden /ID# 34205, Minden
  - Boss, Minden, DE /ID# 145772, Minden
  - Kantner, Moenchengladbach, DE /ID# 99836, Mönchengladbach
  - Zentbeauty Gbr /ID# 72020, Mönchengladbach
  - Stroemer & Deden /ID# 48502, Mönchengladbach
  - Dorittke & Kardorff /ID# 35289, Mönchengladbach
  - Husemann & Fischer, Munich, DE /ID# 53692, Munich
  - Malmusi, Munich, DE /ID# 48450, Munich
  - Anders-Ankerhold, Munich, DE /ID# 53682, Munich
  - Klinikum recht der Isar der TU /ID# 138208, Munich
  - Pfannenstiel, Munich, DE /ID# 126023, Munich
  - TU Uniklinik Munchen /ID# 202198, Munich
  - Gagel, Munich, DE /ID# 60593, Munich
  - Keilig, Munich, DE /ID# 53702, Munich
  - Quack, Munich, DE /ID# 53715, Munich
  - Mang, Muehlhausen, DE /ID# 48451, Mühlhausen
  - Kaufmann, Muehlheim, DE /ID# 60603, Mühlheim
  - Nikodem-Koczwara, Muelheim, DE /ID# 53710, Mülheim
  - Schueller, Muelheim a.d. Ruhr /ID# 126025, Mülheim
  - Habenicht/Marth, Muenster, DE /ID# 138190, Münster
  - Mueller, Muenster, DE /ID# 53709, Münster
  - Lissner, Auerbach, DE /ID# 35061, Münster
  - Wilhelm, Naumburg, DE /ID# 67970, Naumburg
  - Paech, Neubrandenburg, DE /ID# 34057, Neubrandenburg
  - Bruckbauer, Neufahrn, DE /ID# 48418, Neufahrn
  - Franke, Neugersdorf, DE /ID# 138187, Neugersdorf
  - Meisel-Stosiek, Neumarkt, DE /ID# 34067, Neumarkt
  - Schwerbrock, Neumarkt, DE /ID# 34068, Neumarkt
  - Buettner & Meewes,Neumuenster /ID# 35310, Neumünster
  - von Kobyletzki, Nuernberg, DE /ID# 35315, Neustadt
  - Sperling, Neustrelitz, DE /ID# 53721, Neustrelitz
  - Kloos & Loeser, Neuwied, DE /ID# 35318, Neuwied
  - Kloos & Loeser, Neuwied, DE /ID# 35319, Neuwied
  - Boeckers, Nieder-Olm, DE /ID# 138262, Nieder-Olm
  - Mahlke, Norden, DE /ID# 99840, Norden
  - Krankenhaus Norderney /ID# 72021, Norderney
  - Praxis S. Zajac /ID# 148245, Norderstedt
  - Gutgesell, Norderstedt, DE /ID# 34159, Norderstedt
  - Niemeyer, Nordhausen, DE /ID# 35323, Nordhausen
  - Wienrich, Nordhausen, DE /ID# 126029, Nordhausen
  - Thuencher, Nuremberg, DE /ID# 34163, Nuremberg
  - Voelkel, Nuremberg, DE /ID# 34164, Nuremberg
  - Tuerk, Nuremberg, DE /ID# 67968, Nuremberg
  - Praxis Dr.S.Vogel- Kiener /ID# 167679, Nuremberg
  - Vogel/Walther, Nuremberg, DE /ID# 67969, Nuremberg
  - Alpagut & Alpagut & Meisel /ID# 35325, Nuremberg
  - HELIOS St. Elisabeth Klinik /ID# 138263, Oberhausen
  - Saleh, Oberhausen, DE /ID# 138201, Oberhausen
  - Rudolphi/Duckheim, Oberhausen, /ID# 34169, Oberhausen
  - Ponce de Poeschl, Oberschleiss /ID# 53714, Oberschleißheim
  - Hockmann, Oelde, DE /ID# 48515, Oelde
  - Wendrock-Shiga, Oelsnitz, DE /ID# 35328, Oelsnitz
  - Altmeyer, Oer-Erkenschwick, DE /ID# 50783, Oer-Erkenschwick
  - Praxis Dr. Spreng /ID# 145780, Offenbach
  - Fechner/Addicks, Oldenburg, DE /ID# 60582, Oldenburg
  - Reinicke, Oldenburg, DE /ID# 126024, Oldenburg
  - Klinikum Oldenburg GmbH /ID# 50848, Oldenburg
  - Klinikum Oldenburg GmbH /ID# 50854, Oldenburg
  - MVZ Olpe I /ID# 167678, Olpe
  - Reipen, Olpe, DE /ID# 48524, Olpe
  - Fachklinik Bad Bentheim /ID# 35568, Ormond Beach
  - Praxis C. Bochenek /ID# 167671, Oschatz
  - Breitsprecher, Osnabrueck, DE /ID# 35330, Osnabrück
  - Klinikum Osnabrueck GmbH /ID# 35332, Osnabrück
  - Rosenbach, Osnabrueck, DE /ID# 33497, Osnabrück
  - Hoppe, Pasewalk, DE /ID# 53699, Pasewalk
  - Kuehn, Peitz, DE /ID# 33510, Peitz
  - Baumann, Philippsburg, DE /ID# 33518, Philippsburg
  - Staender, Bad Bentheim, DE /ID# 35522, Phoenix
  - Itschert, Pinneberg, DE /ID# 67958, Pinneberg
  - Schmidt, Pirna, DE /ID# 48525, Pirna
  - Kallweit, Plettenberg, DE /ID# 53701, Plettenberg
  - Farzar/Kramer/Mohme, Porta /ID# 33530, Porta Westfalica
  - Farzar/Kramer/Mohme, Porta /ID# 99845, Porta Westfalica
  - Buehler/Radke, Potsdam, DE /ID# 33531, Potsdam
  - Hautarztpraxis am Stadthaus /ID# 141997, Potsdam
  - Hautarztpraxis am Stadthaus /ID# 149287, Potsdam
  - Asadullah/Gross, Potsdam, DE /ID# 72014, Potsdam
  - Luedcke, Potsdam, DE /ID# 33462, Potsdam
  - Praxis Dr. Barbu /ID# 156481, Potsdam
  - MARE Klinikum /ID# 33473, Preetz
  - Akst, Pruem, DE /ID# 33477, Prüm
  - Kirchesch, Pulheim, DE /ID# 50830, Pulheim
  - John&Rupp-John, Puettlingen,DE /ID# 35342, Püttlingen
  - Klin Christiane Erxleben GmbH /ID# 35344, Quedlinburg
  - Frank/Frank, Radebeul, DE /ID# 138186, Radebeul
  - Rozsondai, Radolfzell, DE /ID# 50857, Radolfzell
  - Gehse, Rastatt, DE /ID# 67956, Rastatt
  - Parker, Rastatt, DE /ID# 48522, Rastatt
  - Praxis Dres. Pierchalla & Part /ID# 151478, Recklinghausen
  - Klinikum Univ Regensburg /ID# 33894, Regensburg
  - Haueisen, Regensburg, DE /ID# 81296, Regensburg
  - Kluge & Ott, Rehau, DE /ID# 33895, Rehau
  - Weis, Reichenbach, DE /ID# 138204, Reichenbach
  - Kramer/Mortazawi, Remscheid /ID# 33898, Remscheid
  - Haut-und Allergie-Ambulatorium /ID# 148250, Rendsburg
  - Montag, Rheinbach, DE /ID# 99846, Rheinbach
  - Ludwig, Rheine, DE /ID# 50846, Rheine
  - Manuel, Rheinstetten, DE /ID# 33908, Rheinstetten
  - Maslen & Pavlovsky, Ribnitz /ID# 35353, Ribnitz-Damgarten
  - Krausse, Riesa, DE /ID# 35357, Riesa
  - Krausch, Rinteln, DE /ID# 48447, Rinteln
  - Kleditzsch/Blank, Rostock, DE /ID# 60587, Rostock
  - Buttler, Rostock, DE /ID# 60590, Rostock
  - Hoene, Rostock, DE /ID# 48516, Rostock
  - Slucka, Rostock, DE /ID# 126026, Rostock
  - Goeldner, Rostock, DE /ID# 33919, Rostock
  - Bomke, Rostock, DE /ID# 99816, Rostock
  - Eisfelder, Rottweil, DE /ID# 34010, Rottweil
  - Prifert, Rudolstadt, DE /ID# 35359, Rudolstadt
  - Zapf, Rudolstadt, DE /ID# 34011, Rudolstadt
  - Hempel, Saalfeld, DE /ID# 34013, Saalfeld
  - Trennheuser % Hasselmann /ID# 34018, Saarlouis
  - Salzmann, St. Wendel, DE /ID# 33579, Saint Wendel
  - Spitzbarth, Sangerhausen, DE /ID# 34028, Sangerhausen
  - Broening, Schleiz, DE /ID# 35366, Schleiz
  - Durrant-Finn, Schmoelln, DE /ID# 67950, Schmölln
  - Alscher, Schneeberg, DE /ID# 35368, Schneeberg
  - Gueldner, Schorndorf, DE /ID# 33536, Schorndorf
  - Frankerl, Schwandorf, DE /ID# 33543, Schwandorf in Bayern
  - Mueller, Schwarzenberg, DE /ID# 138197, Schwarzenberg
  - Asklepios Klin Uckermark /ID# 35373, Schwedt
  - Huyke, Schweina, DE /ID# 138193, Schweina
  - Mehringer, Schweinfurt, DE /ID# 50850, Schweinfurt
  - Fraenken/Leksa, Schwelm, DE /ID# 33547, Schwelm
  - von Kiedrowski, Selters, DE /ID# 33560, Selters
  - David, Siegen, DE /ID# 148242, Siegen
  - David, Siegen, DE /ID# 99817, Siegen
  - Asefi, Simmern, DE /ID# 67945, Simmern
  - Albig, Singen, DE /ID# 33564, Singen
  - Hagemann, Soest, DE /ID# 48514, Soest
  - Karl, Soest, DE /ID# 33569, Soest
  - Thiele, Soest, DE /ID# 33568, Soest
  - Wendler, Soemmerda, DE /ID# 138205, Sömmerda
  - Wroblewska, Spaichingen, DE /ID# 34867, Spaichingen
  - Zobel, Spremberg, DE /ID# 50869, Spremberg
  - Blecher, Starnberg, DE /ID# 33589, Starnberg
  - Bange, Stassfurt, DE /ID# 48510, Staßfurt
  - Steinborn, Straubing, DE /ID# 33594, Straubing
  - Cavcic, Stuttgart, DE /ID# 126015, Stuttgart
  - Leitz, Stuttgart, DE /ID# 126018, Stuttgart
  - Leitz, Stuttgart, DE /ID# 72023, Stuttgart
  - Bauer, Stuttgart, DE /ID# 53683, Stuttgart
  - Flegl MD Stuttgart Germany /ID# 50824, Stuttgart
  - Praxis. Dr. Koehler /ID# 142000, Suhl
  - Jager/Landwehr, Sulzbach, DE /ID# 33615, Sulzbach
  - Krusche&Mai,Sulzbach-Rosenberg /ID# 33616, Sulzbach-Rosenberg
  - Kirchhoff, Telgte, DE /ID# 50831, Telgte
  - Lueg, Teltow, DE /ID# 33617, Teltow
  - Cyrulies, Teterow, DE /ID# 33621, Teterow
  - Frank, Tirschenreuth, DE /ID# 33622, Tirschenreuth
  - Meyer, Tornesch, DE /ID# 33626, Tornesch
  - Pleier/Weidenbach, Traunstein, /ID# 33627, Traunstein
  - Brisch, Trier, DE /ID# 60589, Trier
  - Universitatsklinikum Tubingen /ID# 33631, Tübingen
  - Universitatsklinikum Tubingen /ID# 81278, Tübingen
  - Winkler-Gyulay, Unna, DE /ID# 48528, Unna
  - Braun, Ueberlingen, DE /ID# 33638, Überlingen
  - Giesenberg, Varel, DE /ID# 33728, Varel
  - Loetzsch, Varel, DE /ID# 50845, Varel
  - Jasnoch/Kock/Borrosch, Vechta, /ID# 145770, Vechta
  - Jasnoch/Kock/Borrosch, Vechta, /ID# 33730, Vechta
  - Jasnoch/Kock/Borrosch, Vechta, /ID# 60605, Vechta
  - Steiner, Viersen, DE /ID# 141547, Viersen
  - Steiner, Viersen, DE /ID# 99848, Viersen
  - Praxis Dr. Czech /ID# 145765, Villingen-Schwenningen
  - Fischer, Vilshofen, DE /ID# 148252, Vilshofen
  - Fischer, Vilshofen, DE /ID# 50823, Vilshofen
  - Foss, Wadern, DE /ID# 33738, Wadern
  - Barnikol, Waltershausen, DE /ID# 35401, Waltershausen
  - Funke, Waltrop, DE /ID# 33739, Waltrop
  - Hoos, Wedel, DE /ID# 33745, Wedel
  - Billmann-Krutmann, Wegberg, DE /ID# 90958, Wegberg
  - Pausch, Weiden, DE /ID# 60606, Weiden
  - Reindl, Weimar, DE /ID# 60607, Weimar
  - Asklepios Krankenh Weissenfels /ID# 138206, Weißenfels
  - Fiedler, Weissenfels, DE /ID# 33752, Weißenfels
  - Pfennig, Werdau, DE /ID# 48459, Werdau
  - Roehrborn, Werl, DE /ID# 33754, Werl
  - Dr. Barbara Kempkes, Werne /ID# 118540, Werne
  - Jansen & Weersch, Wesel, DE /ID# 33756, Wesel
  - Schmeel, Wesseling, DE /ID# 81303, Wesseling
  - Uszynska-Jast, Wetter, DE /ID# 33758, Wetter
  - Kaempfer, Wetzlar, DE /ID# 33759, Wetzlar
  - Paul, Wetzlar, DE /ID# 50855, Wetzlar
  - Moeller, Wiesbaden, DE /ID# 50852, Wiesbaden
  - Hasselbusch, Wiesmoor, DE /ID# 33766, Wiesmoor
  - Buttgereit/Stiller, Wildau, DE /ID# 33767, Wildau
  - Hutschenreuther, Wilhelmshaven /ID# 33768, Wilhelmshaven
  - Gajda, Wilhelmshaven, DE /ID# 138261, Wilhelmshaven
  - Maronde, Winsen, DE /ID# 53707, Winsen
  - Dr. Martin Gruener, Wipperfuer /ID# 118538, Wipperfürth
  - Klein, Witten, DE /ID# 33777, Witten
  - Hoffmann, Witten, DE /ID# 35417, Witten
  - Merk, Lutherstadt Wittenberg, /ID# 126020, Wittenberg
  - Suess, Wittlich, Germany /ID# 33629, Wittlich
  - Roos, Wittmund, DE /ID# 118542, Wittmund
  - Metz, Wittstock, DE /ID# 33781, Wittstock
  - Franz, Wolfenbuettel, DE /ID# 33782, Wolfenbüttel
  - Rowold, Wolfenbuettel, DE /ID# 48467, Wolfenbüttel
  - Rinke, Wolmirstedt, DE /ID# 48532, Wolmirstedt
  - Fuge-Dierking, Wuppertal, DE /ID# 33720, Wuppertal
  - Gleissner/Sadlo, Wuppertal, DE /ID# 108919, Wuppertal
  - Gleissner/Sadlo, Wuppertal, DE /ID# 48434, Wuppertal
  - Huebinger, Wuppertal, DE /ID# 53700, Wuppertal
  - Praxis Dr. Schock-Skasa /ID# 148246, Wuppertal
  - Bartenberg, Wuppertal, DE /ID# 81273, Wuppertal
  - Albrecht, Wurzen, DE /ID# 35422, Wurzen
  - Beilner-Tack, Wuerzburg, DE /ID# 67947, Würzburg
  - Schubert&Frank&Konrad&Eggert /ID# 33715, Würzburg
  - Schubert&Frank&Konrad&Eggert /ID# 48526, Würzburg
  - Schubert&Frank&Konrad&Eggert /ID# 67961, Würzburg
  - Hamm & Kinkelin, Wuerzburg, DE /ID# 33714, Würzburg
  - Franz-Reichel, Zehdenick, DE /ID# 33860, Zehdenick
  - Weber, Zeulenroda, DE /ID# 50867, Zeulenroda
  - Rudolph, Zschopau, DE /ID# 166129, Zschopau
  - Rudolph, Zschopau, DE /ID# 35424, Zschopau
  - Mischke, Zwickau, DE /ID# 35430, Zwickau
  - Heinrich Braun Klinik Zwickau /ID# 50849, Zwickau
  - Mende-Dietz, Zwickau, DE /ID# 35426, Zwickau
  - Praxis MVZ Gefaesszentrum Zwic /ID# 145766, Zwickau
  - Gebhardt, Zwickau, DE /ID# 35432, Zwickau
  - Junghaenel, Zwickau, DE /ID# 35428, Zwickau

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/clinical-trials/adalimumab_P10-446.pdf